CLINICAL TRIAL: NCT02882685
Title: Comparison of Two Operative Techniques - Mini Gastric Bypass and Roux-en-Y Gastric Bypass in the Treatment of Severe Obesity
Brief Title: Comparison of Mini Gastric Bypass and Roux-en-Y Gastric Bypass
Acronym: RYSA
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Helsinki University Central Hospital (Other)
Responsible Party: Principal Investigator, Tuure Saarinen, MD, Helsinki University Central Hospital
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: HUS214/2016
Record Dates: First submitted 2016-07-23; First posted 2016-08-30 (Estimated); Last update posted 2022-07-20 (Actual); Status verified 2022-07

CONDITIONS: Morbid Obesity
Keywords: Roux-en-Y gastric bypass; Mini-gastric bypass; Single anastomosis gastric bypass
MeSH Terms: conditions — Obesity, Morbid | interventions — Gastric Bypass

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- RYGB (Active Comparator): Roux-en-Y gastric bypass
  Interventions: Procedure: Roux-en-y gastric bypass
- SAGB (Active Comparator): Single anastomosis gastric bypass
  Interventions: Procedure: Single anastomosis gastric bypass

INTERVENTIONS:
Procedure: Roux-en-y gastric bypass
  Other Names: RYGB
  Arms: RYGB
Procedure: Single anastomosis gastric bypass
  Other Names: SAGB; Mini-gastric bypass; MGB
  Arms: SAGB

SUMMARY:
This study compares Roux-en-Y gastric bypass with single anastomosis gastric bypass in a randomized prospective setting. This study also adresses the issue of bile reflux after MGB.

DETAILED DESCRIPTION:
Roux-en-Y gastric bypass (RYGB) and single anastomosis gastric bypass (SAGB or mini gastric bypass, MGB) have both shown excellent weight-loss and effect on comorbidities such as type 2 diabetes.

In this study eligible patients are randomized for either of the operations. Effects on glucose homeostasis as well as weight-loss and the effect on comorbidities are recorded during the follow-up.

Before the surgery and at 6 and 12 months, all participants will undergo body composition measurements (bioimpedance, MRI and DEXA), mixed meal tests and oral glucose tolerance tests, calorimetry and biopsies of skin, subcutaneous fat and muscle will be obtained and samples of urine, feces and saliva are collected. At these timepoints, all patients will fill out questionnaires regarding psychocological, social and physical health and wellbeing.

Interim analysies will be done for the first 60 patients (30 per group) after 3 months, in which safety issues and trial setup is reviewed. If there are no problems with safety and setup, the trial can be carried out according to initial plan.

At 12 months, all outcomes for all patients will be analyzed. Main outcome is weight-loss one year after the surgery.

Follow-up continues at 24months, 5 years and 10 years after the surgery and follow-up data will be analyzed accordingly.

Also, MGB has been feared to cause bile reflux. The first 30 MGB patients will undergo a gastroscopy and a hepatobiliary scintigraphy for bile reflux detection at 6 months.

ELIGIBILITY:
Inclusion Criteria:

* BMI>35

Exclusion Criteria:

* Pregnancy
* Previous bariatric surgery
* Anemia
* esophagitis (LA B-D)
* esophageal intestinal metaplasia

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 120 (Actual)
Dates: Start 2016-07; Primary Completion 2022-12 (Estimated); Study Completion 2026-12 (Estimated)

PRIMARY OUTCOMES:
Weight-loss | One year
  Main outcome is weight-loss at 1 yewar after the operationoperation. Weight-loss is calculated as excess weight-loss compared to the preoperative weight 2 months before the operation.

SECONDARY OUTCOMES:
Glucose homeostasis | Up to 12 months
  2 months before the operation glucose homeostasis status is studied (oral glucose tolerance test). Oral glucose tolerance tests will be repeated at 6months and 12 months. Continuos glucose monitoring will be done before the operation at operation and 6 months after the operation
Bile reflux after Mini Gastric Bypass | 6 months
  All patients undergo a gastroscopy prior to inclusion. Patients with Barrets esophagus or LA B-C esophagitis are excluded. The first 30 patients, who are randomized to Mini Gastric Bypass will undergo a gastroscopy and a hepatobiliary scintigraphy 6 months after the operation. At hepatobiliary scintigraphy the amount of bile reflux is calculated as the amount of tracer found in the gastric pouch or esophagus in relation to total amount of tracer in the liver.
Weight-loss | 10 years
  Weight-loss at 2years, 5years and 10 years

CONTACTS AND LOCATIONS:
Overall Officials: Tuure T Saarinen, MD, Principal Investigator — Helsinki University Central Hospital
Locations (2):
- Finland (2):
  - Helsinki University Central Hospital, Helsinki
  - Oulu University Hospital, Oulu

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] van der Kolk BW, Heinonen S, White JW, Wagner A, Karppinen JE, Saari S, Muniandy M, Metsikko S, Dillon ET, Groop PH, Saarinen T, Le Roux CW, Virtanen KA, Docherty NG, Pirinen E, Juuti A, Pietilainen KH. Human Skeletal Muscle Mitochondria Responses to Weight Loss Induced by Bariatric Surgery or Lifestyle Intervention. Acta Physiol (Oxf). 2026 Feb;242(2):e70150. doi: 10.1111/apha.70150. PMID 41507695
- [Derived] Saarinen T, Merilainen S, Koivukangas V, Pietilainen KH, Juuti A. Prospective randomized controlled trial comparing the efficacy and safety of Roux-en-Y gastric bypass and one-anastomosis gastric bypass (the RYSA trial): trial protocol and interim analysis. Trials. 2019 Dec 30;20(1):803. doi: 10.1186/s13063-019-3898-y. PMID 31888729
- [Derived] Saarinen T, Pietilainen KH, Loimaala A, Ihalainen T, Sammalkorpi H, Penttila A, Juuti A. Bile Reflux is a Common Finding in the Gastric Pouch After One Anastomosis Gastric Bypass. Obes Surg. 2020 Mar;30(3):875-881. doi: 10.1007/s11695-019-04353-x. PMID 31853864